CLINICAL TRIAL: NCT02609698
Title: A Comparative Evaluation of Efficacy and Safety in the 3-Months DAPT Group vs. the 6-Months DAPT Group of Patients Treated With the Coroflex ISAR Stent; A Prospective, Multicenter, Randomized, Open-Label Clinical Trial
Brief Title: ISAR-DAPT (A Comparative Evaluation of Efficacy and Safety in the 3-Months DAPT Group vs. the 6-Months DAPT Group of Patients Treated With the Coroflex ISAR Stent; A Prospective, Multicenter, Randomized, Open-Label Clinical Trial)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: B. Braun Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Myeong-Ho Yoon, Professor, Dept of Cardiology, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJOU-CV-0001
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Stable Angina, Unstable Angina, Silent Coronary Ischemia, Coronary Artery Disease
Keywords: Stent; Polymer-free; Antiplatelet therapy; Clopidogrel; DES; DAPT
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Aspirin; Clopidogrel

ARMS (2):
- Coroflex ISAR 3 months DAPT (Experimental): Patients who have received a Coroflex ISAR stent procedure to treat coronary arterial lesions, and administered the drug for 3 months
  Interventions: Device: Coroflex ISAR; Drug: 3 months DAPT
- Coroflex ISAR 6 months DAPT (Active Comparator): Patients who have received a Coroflex ISAR stent procedure to treat coronary arterial lesions, and administered the drug for 6 months
  Interventions: Device: Coroflex ISAR; Drug: 6 months DAPT

INTERVENTIONS:
Device: Coroflex ISAR — This stent platform has a thin-strut cobalt-chromiun alloy backbone, no polymer, microporous surface.
Drug: 3 months DAPT
  Other Names: Aspirin + clopidogrel for 3-months schedule after the coronary stenting
  Arms: Coroflex ISAR 3 months DAPT
Drug: 6 months DAPT
  Other Names: Aspirin + clopidogrel for 6-months schedule after the coronary stenting
  Arms: Coroflex ISAR 6 months DAPT

SUMMARY:
This clinical trial studies patients treated with the Coroflex ISAR Stent for coronary artery disease in order for the objective of verifying the non-inferiority of results that among patients who were administered DAPT for 3 months compared to patients who were administered DAPT for 6 months, in terms of the efficacy and safety of DAPT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 or older
2. Patients who have submitted a written consent to participate in the clinical trial
3. De novo lesion
4. Patients scheduled for elective intervention to treat ischemic cardiovascular disease

Exclusion Criteria:

1. Patients with any contraindications or hypersensitivity related to antiplatelet therapy
2. Patients with Acute Myocardial Infarction (ST elevation myocardial infarction, Non ST elevation myocardial infarction)
3. Patients who are anticipated to receive treatment or surgery that may require desisting the administration of antiplatelet therapy for 2 weeks or longer during the period of the clinical trial
4. Chronic total occlusion (CTO) lesions, in-stent restenosis (ISR)
5. Patients experiencing cardiogenic shock
6. Women who are breastfeeding, pregnant, or desiring pregnancy
7. Patients with findings of hemorrhage
8. Patients with a life expectancy of less than 1 year
9. Patients who have received a drug-eluting stent (DES) procedure within the past 6 months
10. Any other patients judged by the investigator to be unsuitable for the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 906 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months from the time of the stenting
  Major Adverse Cardiac Events (MACE) (cardiac death, recurrent myocardial infarction, target lesion revascularization) at 12 months from the time of the procedure

SECONDARY OUTCOMES:
MACE | 6 months from the time of the stenting
Any death, cardiac death, MI, TLR, TVR | 6 months from the time of the stenting
Any death, cardiac death, MI, Stroke, TLR, TVR | 12 months from the time of the stenting

CONTACTS AND LOCATIONS:
Overall Officials: Myeong-Ho Yoon, Ph.D, MD, Principal Investigator — Cardiovascular Center, Ajou University Hospital
Locations (1):
- Ajou University Hospital, Yeongtong-gu, Suwon, South Korea

REFERENCES:
- [Derived] Jin U, Seo KW, Yang HM, Lim HS, Choi BJ, Choi SY, Shin JH, Tahk SJ, Yoo SY, Rha SW, Chung WY, Kim CH, Won KB, Pyun WB, Jang JS, Lee SY, Hong YJ, Kim MH, Hong SJ, Choi YS, Kim HY, Choi RK, Kang WC, Cho EJ, Yoon MH. Efficacy and Safety of 3 Versus 6 Months of Dual-Antiplatelet Therapy in Patients Implanted With a Coroflex ISAR Stents: A Prospective, Multicenter, Randomized Clinical Trial. J Invasive Cardiol. 2022 Sep;34(9):E653-E659. doi: 10.25270/jic/21.00330. Epub 2022 Jul 22. PMID 35863061